CLINICAL TRIAL: NCT07348835
Title: Continuous Monitoring Using a Smart Implantable Device (Persona IQ®) to Compare Medial Parapatellar vs. Subvastus Approaches in Early Post-Operative Total Knee Arthroplasty Recovery
Brief Title: Using a Smart Implantable Device to Compare Early Recovery in Two Different Knee Arthroplasty Approaches
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Total Joint Specialists (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSH1432
Record Dates: First submitted 2025-12-15; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Total Knee Anthroplasty
Keywords: Total Knee Arthroplasty; Medial Parapatellar Approach; Subvastus Approach

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, parallel-group study. Eligible patients undergoing primary total knee arthroplasty are randomized in a 1:1 ratio to either the medial parapatellar or subvastus surgical approach and followed concurrently. Outcomes are assessed longitudinally.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medial Parapatellar Approach (Active Comparator): Primary total knee arthroplasty performed using the medial parapatellar surgical approach
  Interventions: Procedure: Total Knee Arthroplasty Medial Parapatellar Approach
- Subvastus Approach (Active Comparator): Primary total knee arthroplasty performed using the subvastus surgical approach
  Interventions: Procedure: Total Knee Arthroplasty Subvastus Approach

INTERVENTIONS:
Procedure: Total Knee Arthroplasty Medial Parapatellar Approach — Incision splitting quad
  Arms: Medial Parapatellar Approach
Procedure: Total Knee Arthroplasty Subvastus Approach — quad-sparing approach
  Arms: Subvastus Approach

SUMMARY:
This is a single-institution, prospective, randomized study comparing the medial parapatellar and subvastus approaches in primary total knee arthroplasty using continuous, implant-based gait monitoring. Patients receiving a Zimmer Persona IQ smart implant will be followed preoperatively and through the first 30 days post-operatively, with extended follow-up to 6 months. Preoperative activity is captured using iPhone Health step-count data, while post-operative recovery is assessed using continuous tibial implant data, including step count, range of motion, cadence, walking speed, stride length, and distance. These objective metrics are correlated with PROMs. The primary outcome is daily step count. Secondary outcomes include early functional milestones, pain, and patient-reported functional scores. This study is designed to characterize early recovery trajectories and determine whether meaningful differences exist between surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years of age who plan to undergo medial congruent polyethylene bearing primary TKA with a PIQ
* Eligible for both approaches
* Have an iPhone and willing to "wear" it for two weeks preoperatively to get an estimated average stepcount
* Provide informed consent
* Willing to complete follow ups

Exclusion Criteria:

* Patients with TKA revisions
* Patients with insufficient pre-operative range of motion in the operative knee (flexion contracture of > 20 degrees or < 90° of knee flexion)
* Patients with Contralateral TKA within study time frame
* Patients with TKA other than medial congruent polyethylene bearing
* Patients with bilateral surgery
* Patients without a valid and active email address
* Patients not willing or able to participate in study and follow-ups
* Patients who use assisted devices to ambulate
* Rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Step Count (steps/day) | Through study completion, minimum 6 months
  Continuously recorded from PIQ device after it is implanted during surgery
Step Count (steps/day) | Baseline
  Recorded from patients iPhone Health App for 2 weeks preoperatively

SECONDARY OUTCOMES:
Stride Length (m) | Through study completion, minimum 6 months
  Continuously recorded from PIQ device after it is implanted during surgery
Distance Travelled (km) | Through study completion, minimum 6 months
  Continuously recorded from PIQ device after it is implanted during surgery
Functional Range of Motion (degrees) | Through study completion, minimum 6 months
  Continuously recorded from PIQ device after it is implanted during surgery
Tibial Range of Motion (degrees) | Through study completion, minimum 6 months
  Continuously recorded from PIQ device after it is implanted during surgery
Cadence (steps/minute) | Through study completion, minimum 6 months
  Continuously recorded from PIQ device after it is implanted during surgery
Walking Speed (m/s) | Through study completion, minimum 6 months
  Continuously recorded from PIQ device after it is implanted during surgery
Goniometric Functional Range of Motion | Preoperatively and at 6 weeks
  Measured in degrees using a goniometer
Surgical Side | Preoperatively
  Left or Right
Age | Preoperatively
  In years, from EMR
Sex | Preoperatively
  Male or Female, from EMR
Weight | Preoperatively
  In kg, from EMR
Height | Preoperatively
  In cm, from EMR
Body Mass Index (BMI) | Preoperatively
  in kg/m2, from EMR
Comorbidities | Preoperatively
  Collected and listed from EMR
Charlson Comorbidity Index (CCI) | Preoperatively
  Calculated from formula using comorbidities collected from EMR
Time to Achieving Key Milestones in Daily Activities | 6 weeks postoperatively
  Survey score collected (less time = better), Survey via Force Therapeutics
Veterans Rand 12-Item (VR-12) Health Survey | Preoperatively, 6 weeks postoperatively, 6 months postoperatively
  Mental and Physical component survey scores collected (0-100); Survey via Force Therapeutics
Procedure Satisfaction | 6 weeks postoperatively
  Survey score collected (0-5; 5 best), Survey via Force Therapeutics
Numeric Pain Rating Scale (NPRS) | Preoperatively, 6 weeks postoperatively
  Survey score collected (0-10; 0 best), Survey via Force Therapeutics
Knee injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR.) | Preoperatively, 6 weeks postoperatively, 6 months postoperatively
  Survey score collected (0-100; 100 best), Survey via Force Therapeutics
Forgotten Joint Score (FJS) | Preoperatively, 6 weeks postoperatively, 6 months postoperatively
  Survey score collected (0-100; 100 best), Survey via Force Therapeutics

CONTACTS AND LOCATIONS:
Locations (1):
- Total Joint Surgery Center Atlanta, Sandy Springs, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be used as necessary by the authorized research team and always secured, it will not be shared

REFERENCES:
- [Background] Matsueda M, Gustilo RB. Subvastus and medial parapatellar approaches in total knee arthroplasty. Clin Orthop Relat Res. 2000 Feb;(371):161-8. doi: 10.1097/00003086-200002000-00020. PMID 10693563
- [Background] Kazarian GS, Siow MY, Chen AF, Deirmengian CA. Comparison of Quadriceps-Sparing and Medial Parapatellar Approaches in Total Knee Arthroplasty: A Meta-Analysis of Randomized Controlled Trials. J Arthroplasty. 2018 Jan;33(1):277-283. doi: 10.1016/j.arth.2017.08.025. Epub 2017 Aug 30. PMID 28947369
- [Background] Cila E, Guzel V, Ozalay M, Tan J, Simsek SA, Kanatli U, Ozturk A. Subvastus versus medial parapatellar approach in total knee arthroplasty. Arch Orthop Trauma Surg. 2002 Mar;122(2):65-8. doi: 10.1007/s004020100319. PMID 11880904
- [Background] Tomek IM, Kantor SR, Cori LA, Scoville JM, Grove MR, Morgan TS, Swarup I, Moschetti WE, Spratt KF. Early Patient Outcomes After Primary Total Knee Arthroplasty with Quadriceps-Sparing Subvastus and Medial Parapatellar Techniques: A Randomized, Double-Blind Clinical Trial. J Bone Joint Surg Am. 2014 Jun 4;96(11):907-915. doi: 10.2106/JBJS.L.01578. Epub 2014 Jun 4. PMID 24897738
- [Background] Sukeik M, Sohail MZ, Hossain FS, AlShryda S, Powell J. Comparing the Sub-Vastus and Medial Parapatellar Approaches in Total Knee Arthroplasty: A Meta-Analysis of Short-Term Outcomes. Dr Sulaiman Al Habib Med J. 2021;3(2):66. doi:10.2991/dsahmj.k.210203.001
- [Background] Khan MNH, Abbas K, Faraz A, Ilyas MW, Shafique H, Jamshed MH, Hashmi P. Total knee replacement: A comparison of the subvastus and medial parapatellar approaches. Ann Med Surg (Lond). 2021 Aug 8;68:102670. doi: 10.1016/j.amsu.2021.102670. eCollection 2021 Aug. PMID 34408867
- [Background] van Hemert WL, Senden R, Grimm B, van der Linde MJ, Lataster A, Heyligers IC. Early functional outcome after subvastus or parapatellar approach in knee arthroplasty is comparable. Knee Surg Sports Traumatol Arthrosc. 2011 Jun;19(6):943-51. doi: 10.1007/s00167-010-1292-0. Epub 2010 Oct 17. PMID 20953864
- [Background] Ambrosino C, Ubertalle A, Liberatori J, Sarra C. [Proteins of milk sera. VI. Research by microimmunodiffusion in agar gel on immunochemical behavior of the sera of cow, sheep, goat and buffalo milk]. Ric Sci 2 Ser Pt 2 Rend B. 1965 Apr-Jun;6(2):125-34. No abstract available. Italian. PMID 5890136
- See also: Persona IQ Device — https://www.zimmerbiomet.com/en/products-and-solutions/specialties/knee/persona-iq.html

DOCUMENTS (2):
  • Study Protocol (2025-10-31): https://cdn.clinicaltrials.gov/large-docs/35/NCT07348835/Prot_000.pdf
  • Informed Consent Form (2025-10-31): https://cdn.clinicaltrials.gov/large-docs/35/NCT07348835/ICF_001.pdf